CLINICAL TRIAL: NCT02148107
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 691751 in Healthy Male Subjects
Brief Title: Multiple Rising Oral Doses of BI 691751 in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1334.2; 2013-003813-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

ARMS (7):
- BI 691751 Dose 1 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- BI 691751 Dose 2 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- BI 691751 Dose 3 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- BI 691751 Dose 4 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- BI 691751 Dose 5 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- BI 691751 Dose 6 (Experimental): multiple dose given over 14 days
  Interventions: Drug: BI 691751
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 691751 — BI 691751 Dose 1
  Arms: BI 691751 Dose 1
Drug: BI 691751 — BI 691751 Dose 2
  Arms: BI 691751 Dose 2
Drug: BI 691751 — BI 691751 Dose 3
  Arms: BI 691751 Dose 3
Drug: BI 691751 — BI 691751 Dose 4
  Arms: BI 691751 Dose 4
Drug: BI 691751 — BI 691751 Dose 5
  Arms: BI 691751 Dose 5
Drug: BI 691751 — BI 691751 Dose 6
  Arms: BI 691751 Dose 6
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
It is the objective of this MRD trial to investigate pharmacokinetics, pharmcodynamics, safety and tolerability of rising doses BI 691751 over a treatment period of 14 days to support the further clinical development of this LTA4H-inhibitor. Special emphasis will be given to detect potential effects of BI 691751 on heart rate.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator´s assessment, based on a complete medical history including a physical examination, vital signs (BP (blood pressure), PR (pulse rate), 12-lead ECG (electro cardiogramm), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI (body mass index) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP(Good Clinical Practice) and local legislation
* Subject is able to understand and communicate in German

Exclusion criteria:

* Any finding in the medical examination (including BP (blood pressure), PR (pulse rate) or ECG (electro cardiogramm) is deviating from normal and judged as clinically relevant by the investigator
* Pulse rate outside 45-80 bpm (beats per minutes) or repeated measurement of systolic blood pressure greater than 140 mmHg, diastolic blood pressure greater than 90 mm Hg
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication
* Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during inhouse-confinement
* Alcohol abuse (consumption of more 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Vulnerable subjects, e.g. subjects kept in detention, soldiers, employees of the sponsor or a clinical research organization, involved in this study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1334.2.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was terminated early therefore only the first 2 dose levels planned (0.5 mg and 3.0 mg) were administered. In addition, due to recruitment problems fewer subjects than planned were randomised into the placebo and BI 691751 3mg groups.
Groups:
- BI 691751 0.5mg: Oral administration of a BI 691751 0.5mg tablet taken once daily for 14 days
- BI 691751 3mg: Oral administration of BI 681751 3mg, consisting of two 0.5 mg tablets and a 2mg tablet, taken once daily for 14 days.
- Placebo: Oral administration of a placebo tablet matching the BI 691751 tablets, taken once daily for 14 days.
Period: Overall Study
Arm/Group | BI 691751 0.5mg | BI 691751 3mg | Placebo
Started | 8 | 7 | 3
Completed | 8 | 7 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 691751 0.5mg | BI 691751 3mg | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (5.9) | 29.7 (2.8) | 33.3 (2.1) | 32.0 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 7 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related Adverse events (AEs)
Time Frame: From the time of administration of the respective treatment until 21 days after last administration of study drug or start of the post-study phase to the respective treatment, up to 35 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | BI 691751 0.5mg | BI 691751 3mg | Placebo
Number analyzed (Participants) | 8 | 7 | 3
Percentage of participants | 0 | 28.6 | 0

2. Secondary Outcome: AUCt,1 (Area Under the Concentration-time Curve of the Analyte in Plasma Over a Uniform Dosing Interval t After Administration of the First Dose)
Description: AUCt,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose).
  This endpoint could not be calculated as no PK blood samples were analysed due to the early termination of the study.
Time Frame: 0 minutes (min), 10min, 20min, 40min, 1 hour (h), 1h 30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h and 24h after first drug administration
Population: PK set. As no PK blood samples were analysed due to the early termination of the study, no PK parameters could be calculated and so the PK set contains 0 participants.
Arm/Group | BI 691751 0.5mg | BI 691751 3mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cmax (Maximum Measured Concentration of the Analyte Inplasma)
Description: Cmax (maximum measured concentration of the analyte inplasma).
  This endpoint could not be calculated as no PK blood samples were analysed due to the early termination of the study.
Time Frame: as for outcome 2
Population: as for outcome 2
Arm/Group | BI 691751 0.5mg | BI 691751 3mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: AUCt,ss (Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t)
Description: AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t).
  This endpoint could not be calculated as no PK blood samples were analysed due to the early termination of the study.
Time Frame: 312 hours (h), 312 h 10 minutes (min), 312h 20min, 312h 40min, 313, 313h 30min, 314h, 315h, 316h, 318h, 320h, 322h, 324h and 336h after first drug administration
Population: as for outcome 2
Arm/Group | BI 691751 0.5mg | BI 691751 3mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cmax,ss (Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval t)
Description: Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t).
  This endpoint could not be calculated as no PK blood samples were analysed due to the early termination of the study.
Time Frame: as for outcome 4
Population: as for outcome 2
Arm/Group | BI 691751 0.5mg | BI 691751 3mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of administration of the respective treatment until 21 days after last administration of study drug or start of the post-study phase to the respective treatment, up to 35 days
Arm/Group | Placebo | BI 691751 0.5mg | BI 691751 3mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/3 | 2/8 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | BI 691751 0.5mg (N=8) | BI 691751 3mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated prematurely because the sponsor decided to discontinue the development of BI 691751, also no PK blood samples were analysed because of the trial termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.